CLINICAL TRIAL: NCT05547386
Title: 68Ga-PSMA-11 PET/CT for Screening Prior to 177Lu-PSMA-617 Therapy
Brief Title: 68Ga-PSMA-11 PET/CT Screening Prior to 177Lu-PSMA-617 Therapy for Patients With Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Geoffrey Johnson, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-003732; NCI-2022-04135 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Observational (68Ga-PSMA-11 PET/CT) (Experimental): Patients receive 68Ga-PSMA-11 IV and then undergo a PSMA PET/CT scan throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase III study provides access to 68Ga-PSMA-11 positron emission tomography (PET)/computed tomography (CT) imaging for patients with castrate-resistant prostate cancer that has spread to other places in the body (metastatic) being considered for177Lu-PSMA-617 therapy. T PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of this tracer. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. Combining a PET scan with a CT scan can help make the images easier to interpret. The 68Ga-PSMA-11 PET/CT scan is done with a very small amount of radioactive tracer call 68- gallium PSMA-11. In patients that have been diagnosed with prostate cancer, a protein called prostate-specific membrane antigen (PSMA) appears in large amounts on the surface of the cancerous cells. The radioactive imaging agent (68Ga-PSMA-11) has been designed to circulate through the body and attach itself to the PSMA protein on prostate cancer cells. A PET/CT scan is then used to detect the location of prostate cancer lesions. By gaining access to 68Ga-PSMA-11 PET/CT scans, patients may be safely screened for 177Lu-PSMA-617 therapy in the treatment of metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To overcome a clinical access issue that would otherwise block patients from reimbursement of a new cancer therapy, and therefore block or significantly delay their care.

OUTLINE:

Patients receive gallium Ga 68 gozetotide intravenously (IV) and then undergo a positron emission tomography (PET)/computed tomography (CT) scan throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* An adult male patient who is actively under the care of a medical oncology, radiation oncology or urology physician at Mayo Clinic
* An adult male patient who is deemed eligible (or potentially/likely eligible) for PSMA-targeted radionuclide therapy by a nuclear medicine physician or Radiologist in the nuclear medicine therapy practice, or by the Prostate Theranostic Tumor Board (PTuB)

  * Eligibility will be documented in the medical record by the clinical practice
  * It is acceptable for the patient to be eligible for PSMA-targeted radionuclide therapy in all regards except for having completed a PSMA-targeted PET scan showing PSMA-positive prostate cancer
  * It is acceptable for a patient to be potentially eligible for therapy, but have a relative contraindication, such as a minor laboratory abnormality, and be on the list for discussion at the PTuB in the future
* An adult male patient who has not received a 68Ga-PSMA-11 PET/CT or PET/magnetic resonance (MR), or for whom a repeat 68Ga-PSMA-11 PET/CT exam is needed per the clinical practice to ensure eligibility
* An adult male patient who does not otherwise have access to a reimbursable clinical 68Ga-PSMA-11 PET scan
* An adult above the ages of 18

Exclusion Criteria:

* A patient who is unable to consent per Mayo guidelines
* A patient who is unable to lay still, or otherwise successfully complete the imaging exam

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey B. Johnson, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational (68Ga-PSMA-11 PET/CT)
Started | 163
Completed | 156
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Observational (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 163
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 1
  40-49 | 1
  50-59 | 9
  60-69 | 63
  70-79 | 69
  80-89 | 18
  90-99 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 163
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 163

OUTCOME MEASURES:

1. Primary Outcome: Patients Reporting Adverse Reactions
Description: Safety of gallium Ga 68 gozetotide [68Ga-prostate-specific membrane antigen (PSMA)-11] assessed by the number of patients reporting unexpected adverse reactions from the time of injection until the time they leave the care of the division of nuclear medicine. If any adverse reactions are reported, the patient will be evaluated by a nurse and/or physician and will receive appropriate care. The principal investigator (PI) or those designated by the PI will ascertain the severity of the adverse event and how likely the adverse reaction was associated with the injected 68Ga-PSMA-11.
Time Frame: From the time of injection until the time after imaging scan is complete, up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 156
Participants | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for 24 hours after receiving injection/nuclear medicine scans
Arm/Group | Observational (68Ga-PSMA-11 PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156
Other Adverse Events (participants affected / at risk) | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT05547386/Prot_000.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT05547386/ICF_001.pdf